CLINICAL TRIAL: NCT04384146
Title: PROMISE 006: A Phase I Study of up to 3 Cycles of Cyclical Hypofractionated Palliative Radiation (Quad Shot) for Lung Tumors in Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Radiation Therapy to Relieve Symptoms in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-148
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Cyclical Hypofractionated Palliative Radiation (Quad Shot; 20-148
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Phase I, prospective trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Quad Shot Radiation (Experimental): In this trial, patients with centrally located lung tumors will be treated with up to 3 cycles of Quad Shot Radiation. Radiation treatment will be given within 1 week of administration of chemotherapy. Quad Shot radiation will involve: 3.7 Gy twice daily x 2 days for a total dose of 14.8 Gy per cycle. The next cycle will occur after a 21-28 day break. The first group of patients will be treated with 2 cycles of quad shot radiation, followed by a 3-month observation period post-RT to allow a complete evaluation of acute toxicity. The next group of patients will be treated with either 1 cycle or 3 cycles of quad shot radiation. The minimum accrual is 4 patients with an expected accrual of 16 patients. Twenty additional patients will be recruited to an expansion cohort.
  Interventions: Radiation: Cyclical Hypofractionated Palliative Radiation (Quad Shot); Behavioral: EORTC QLQ-C30 questionnaire

INTERVENTIONS:
Radiation: Cyclical Hypofractionated Palliative Radiation (Quad Shot) — 3.7 Gy twice daily x 2 days for a total dose of 14.8 Gy per cycle. The next cycle will occur after a 21-28 day break.
Behavioral: EORTC QLQ-C30 questionnaire — at baseline, each cycle of Quad Shot, and at 3 weeks, 3 months and 6 months after last cycle of Quad Shot.

SUMMARY:
This study will test the safety of Quad Shot radiation therapy using 2 different treatment schedules to find out what effects, if any, this treatment has on people with advanced NSCLC who are receiving systemic therapy for their cancer. The Quad Shot treatment schedule reduces the number of days needed to deliver the radiation treatments, which may be less disruptive to systemic therapy schedules.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer with metastatic disease detected on cross-sectional imaging with a plan for one of the following systemic therapies:

  * Carboplatin/paclitaxel
  * Carboplatin/paclitaxel/pembrolizumab
  * Carboplatin/pemetrexed
  * Carboplatin/pemetrexed/pembrolizumab
  * Pembrolizumab (single agent or in combination with other regimens in this list)
  * Cisplatin/pemetrexed
  * Cisplatin/pemetrexed/pembrolizumab
  * Pemetrexed/pembrolizumab
  * Pemetrexed
  * Nivolumab (single agent or in combination with other regimens in this list)
  * Ipilimumab/nivolumab
  * Carboplatin/etoposide
  * Carboplatin/etoposide/atezolizumab
  * Cisplatin/etoposide
  * Cisplatin/etoposide/atezolizumab
  * Durvalumab (single agent or in combination with other regimens in this list)
  * Atezolizumab (single agent or in combination with other regimens in this list)
* Patients eligible for the systemic therapy regimens notes
* Patients with Stage IV NSCLC who have symptomatic (defined by patient-reported cough, dyspnea, or hemoptysis) or near-symptomatic (determined radiographically to be threatening the airway, esophagus or vasculature) centrally located.
* KPS ≥ 60
* Age ≥ 18 years.
* Able to provide informed consent.
* Patients at reproductive potential must agree to practice an effective contraceptive method.

Exclusion Criteria:

* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances.
* Serious medical co-morbidities precluding radiotherapy.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2026-02-05 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 3 months
  Dose Limiting Toxicity will be defined by CTCAE v5 grade 3 or higher for Esophagitis, Pneumonitis, Bronchial, bronchopleural or tracheal fistula, Bronchopulmonary or mediastinal hemorrhage. Patients will be evaluable for AE/DLTs from the start of study therapy through the end of the 3-month observation period

SECONDARY OUTCOMES:
Number of participants who are able to complete the assigned radiation therapy regimen (3 cycles of quad shot) | 1 year
  To assess the feasibility of delivering up to 3 cycles of quad shot palliative radiation therapy to Stage IV NSCLC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ma, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm